CLINICAL TRIAL: NCT02878629
Title: Mandibular Advancement Devices Tali® in Patients With Syndrome of Obstructive Sleep Apnea and Hypopneas
Status: Completed | Type: Observational
Sponsor: ONIRIS (Industry)
Responsible Party: Sponsor
Other Study IDs: OAM Tali®
Record Dates: First submitted 2016-08-22; First posted 2016-08-25 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Syndrome of Obstructive Sleep Apnea and Hypopneas
MeSH Terms: interventions — Occlusal Splints

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Device: Mandibular Advancement Devices

SUMMARY:
The main objective is to evaluate middle term compliance (≥ 2 years) of the Mandibular Advancement Devices Tali® in patients with Syndrome of Obstructive Sleep Apnea and Hypopneas.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years treated with Mandibular Advancement Device Tali® from at least 2 years and at the latest 5 years.
* Patients who agree to participate to the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients > 18 years treated with Mandibular Advancement Device Tali® from at least 2 years and at the latest 5 years.
Sampling Method: Probability Sample
Enrollment: 254 (Actual)
Dates: Start 2016-07; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
compliance (no stop of the Mandibular Advancement Device) | 2 years or more after the beginning of device

CONTACTS AND LOCATIONS:
Locations (1):
- Liberal cabinet, Paris, France